CLINICAL TRIAL: NCT02366039
Title: Probe-based Volumetric Laser Endomicroscopy (pVLE) of Endoscopic Mucosal Resection (EMR) Tissue in Patients With Barrett's Dysplasia
Acronym: VLE EMR
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Other Study IDs: 12-006665
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Barrett's Esophagus With High Grade Dsyplasia; Early Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMR: patients undergoing clinically indicated endoscopic mucosal resection as standard of care will be asked to participate for this observational study

SUMMARY:
This study is to assess the diagnostic accuracy and precision of the Probe-based Volumetric Laser Endomicroscopy (pVLE) imaging system in detecting dysplasia in BE in both in vivo and ex vivo imaging of Endoscopic Mucosal Resection (EMR) tissue, as compared to standard histopathology

DETAILED DESCRIPTION:
To assess the ability of pVLE to visualize subsurface architecture of EMR tissue, as compared to histology in both in vivo and ex vivo imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females over the age of 18 years.
2. Patients with either suspected or confirmed Barrett's-associated high grade dysplasia (HGD) or intramucosal cancer (IMC) presenting for endoscopy possibly requiring EMR.
3. Ability to provide written, informed consent.
4. Females must be willing to take a pregnancy test if still capable of bearing a child.

Exclusion Criteria:

1. Patients on anticoagulation undergoing high risk procedures in accordance to ASGE guideline for the management of antithrombotic agents for endoscopic procedures (2009)*.
2. Patients with esophageal varices that preclude biopsies.
3. Presence of an esophageal mass/cancer that precludes full distention of the balloon from the Nvision balloon guide sheath.
4. Patients with esophageal strictures that would prevent adequate expansion of the balloon from the Nvision guide sheath.
5. Patients with known inflammatory disease, esophageal tears or ulcers, which prohibit full distention of the balloon from the Nvision balloon guide sheath.
6. Patients with known eosinophilic esophagitis.
7. Patients who are pregnant.
8. Patients with a history of hemostasis disorders*.

   * Patients on anticoagulation undergoing low risk procedures are not excluded. ** Hemostasis disorders will include, but will not be limited to: patients with hemophilia or other congenitally acquired clotting factor deficiencies, patients with cirrhosis with coagulopathy, patients known to have thrombocytopenia (<100,000 plt/ul) and individuals with von Willebrand's disease or other known platelet malfunction disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects undergoing clinically-indicated EMR for BE dysplasia will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-09; Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
distinguishing between normal esophageal squamous mucosa and Barrett's dysplasia | at time of endoscopic mucosal resection
  We will assess descriptive and diagnostic performance (accuracy, sensitivity, specificity, positive and negative predictive values) of the Nvision pVLE device in visualizing dysplasia as compared to standard histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Cadman Leggett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials